CLINICAL TRIAL: NCT06656884
Title: FARAPULSE Workflow Assessment Registry
Acronym: FARAWAY
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PF117
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Catheter Ablation; Pulsed Field Ablation; FARAPULSE; Workflow Assessment
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is designed to determine the best practices in the patient pathway, and to analyze pre-procedural, procedural and follow-up workflow data related with ablation of atrial fibrillation where the FARAPULSE™ Pulsed Field Ablation System is used in a commercial and standard of care setting. Workflow-related variables, inclusive of pre-procedural imaging, methods of transseptal access, anesthesia/sedation technique, intracardiac mapping, ablation settings, dosing strategy, lesion sets and general procedure management, will be used to identify predominant workflow schemes that will be associated with patient demographics, procedure-related complications (safety parameters), and one-year effectiveness parameters.

The study data can be used for procedural workflow optimization when using Pulsed Field Ablation for the ablation treatment of Atrial Fibrillation based on patient demographics, cardiac anatomy and arrhythmia characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are prospectively planned and intended to be treated with the FARAPULSE™ Pulsed Field Ablation system for cardiac tissue ablation, per physician's medical judgement, and as per hospitals' standard of care
* Subjects who are willing and capable of providing informed consent
* Subjects who are willing and capable of participating to this Registry at an approved clinical investigational center
* Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study. Exceptions are when the subject is participating in a mandatory governmental registry, or a purely observational registry, that do not interfere with the current study
* Prior Left Atrium Ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Subjects who will undergo an ablation procedure with the FARAPULSE™ Pulsed Field Ablation system, per physician's medical judgement, and according to hospitals' standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Association of patient demographics with Index procedure Workflow-related variables | Index Procedure
  Patient demographics such as age (years), gender, BMI (kg/m²), different comorbidities, LA Volume (ml), PV anatomy, AF type, pre-procedural AF management) will be compared with different index procedure workflow related variables such as pre-procedural imaging, method and location of transseptal access, intracardiac electro-anatomical mapping, imaging techniques, anesthesia/sedation technique, ablation settings, dosing strategy, lesion sets and general procedure management
Association of safety parameters with Index procedure Workflow-related variables | 12 months
  Safety parameters such as device or procedure related serious adverse events (within 7 days onset date) Death; Myocardial Infarction; Stroke; TIA; Peripheral or Organ Thromboembolism; Pulmonary Edema; Unresolved Phrenic Nerve Palsy/Paresis at 12 Months post-Index Procedure; Vascular Access Complications; Heart Block; Gastric Motility / Pyloric Spasm Disorders, Cardiac Tamponade / Perforation; Pericarditis; Severe Hemolysis with Subsequent Renal Injury or Significant Anemia / Within 12 Months onset date: Pulmonary Vein Stenosis; Atrio-Esophageal Fistula) will be compared with different index procedure workflow related variables such as pre-procedural imaging, method and location of transseptal access, intracardiac electro-anatomical mapping, imaging techniques, anesthesia/sedation technique, ablation settings, dosing strategy, lesion sets and general procedure management
Association of effectiveness parameters with Index procedure Workflow-related variables | 12 months
  Acute and long-term (freedom from AF episodes and freedom from intervention for AF/AFL/AT) Effectiveness parameters will be compared with different index procedure workflow related variables such as pre-procedural imaging, method and location of transseptal access, intracardiac electro-anatomical mapping, imaging techniques, anesthesia/sedation technique, ablation settings, dosing strategy, lesion sets and general procedure management
Association of patient demographics with effectiveness parameters | 12 months
  Patient demographics such as age (years), gender, BMI (kg/m²), different comorbidities, LA Volume (ml), PV anatomy, AF type, pre-procedural AF management) will be compared with Acute and long-term (freedom from AF episodes and freedom from intervention for AF/AFL/AT) Effectiveness parameters
Association of patient demographics with safety parameters | 12 months
  Patient demographics such as age (years), gender, BMI (kg/m²), different comorbidities, LA Volume (ml), PV anatomy, AF type, pre-procedural AF management) will be compared with Safety parameters such as device or procedure related serious adverse events (within 7 days onset date) Death; Myocardial Infarction; Stroke; TIA; Peripheral or Organ Thromboembolism; Pulmonary Edema; Unresolved Phrenic Nerve Palsy/Paresis at 12 Months post-Index Procedure; Vascular Access Complications; Heart Block; Gastric Motility / Pyloric Spasm Disorders, Cardiac Tamponade / Perforation; Pericarditis; Severe Hemolysis with Subsequent Renal Injury or Significant Anemia / Within 12 Months onset date: Pulmonary Vein Stenosis; Atrio-Esophageal Fistula)

CONTACTS AND LOCATIONS:
Locations (33):
- A.o. Krankenhaus der Elisabethinen Linz, Linz, Austria
- Belgium (3):
  - Ziekenhuis aan de Stroom, Middelheim, Antwerp
  - Ziekenhuis Oost-Limburg, Genk
  - CHR de la Citadelle, Namur
- France (3):
  - CHU de Bordeaux, Bordeaux
  - Hopital Saint Philibert, Lomme
  - CHRU Hopital Trousseau, Tours
- Germany (5):
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
  - Munchen Klinik Bogenhausen, München
  - University Hospital of Muenster, Münster
- Greece (2):
  - Ippokrateio General Hospital of Athens, Athens
  - Mitera Hospital, Athens
- Italy (5):
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Ospedale Dell Angelo, Mestre
  - Azienda Ospedaliera San Gerardo, Monza
  - Ospedale di Rivoli, Rivoli
  - Ospedale San Bortolo di Vicenza Azienda ULSS 8 Berica, Vicenza
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands
- King Fahd Armed Forces Hospital, Jeddah, Saudi Arabia
- Spain (4):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - University Hospital Virgen Arrixaca, El Palmar
  - Hospital de Navarra, Pamplona
  - Hospital Universitario Nuestra Senora de Candelaria, Santa Cruz de Tenerife
- GHP Arytmi Center Stockholm, Stockholm, Sweden
- United Kingdom (7):
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - Papworth Hospital, Cambridge
  - Glenfield Hospital, Leicester
  - St. Georges Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Southampton University Hospital, Southampton